CLINICAL TRIAL: NCT04912089
Title: Enhancing Transdiagnostic Mechanisms of Cognitive Dyscontrol Using Computer-based Training
Brief Title: Enhancing Transdiagnostic Mechanisms of Cognitive Dyscontrol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jessica Bomyea, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 210686
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Anxiety Disorders; Depression; Posttraumatic Stress Disorder
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic | interventions — cogent db

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Training Low Dose (Experimental): Cognitive training completed for 8 sessions
  Interventions: Behavioral: COGENT
- Cognitive Training High Dose (Experimental): Cognitive training completed for 16 sessions
  Interventions: Behavioral: COGENT
- Repeat Assessment (No Intervention)

INTERVENTIONS:
Behavioral: COGENT — COGENT is based on a working memory capacity task, which requires individuals to memorize stimuli while simultaneously completing a secondary puzzle task.
  Arms: Cognitive Training High Dose; Cognitive Training Low Dose

SUMMARY:
The proposed project aims to test the cognitive and neural effects of a cognitive training in a sample of individuals seeking treatment for anxiety, depression, or traumatic stress symptoms. Participants will be randomly assigned to a high dose, low dose, or assessment only condition. Participants will be compared on cognitive performance and brain response during cognitive tasks from baseline to post-treatment.

DETAILED DESCRIPTION:
Mood, anxiety, and traumatic stress disorders are common psychiatric conditions - affecting over 40 million U.S. adults - and are leading causes of disability worldwide. People with these conditions are commonly plagued by difficulty controlling distressing personal thoughts and memories, collectively referred to as repetitive negative thinking symptoms. Models suggest that repetitive negative thinking is driven by executive functioning deficits, such that cognitive resources are insufficient to downregulate unwanted thoughts. Executive functioning deficits could be a promising treatment target but are not typically addressed with existing interventions. The long-term goal advanced by this project is to develop effective, mechanistic cognitive training programs that can improve cognition and reduce symptoms associated with mood, anxiety, and traumatic stress disorders. The objectives of this proposal are first to determine the optimal dose of a cognitive training program designed to improve executive functioning in this population using behavioral and neural outcomes. The central hypothesis is that repeated training exercises will enhance executive functioning and will lead to a reduction of repetitive negative thinking in mood, anxiety, and traumatic stress disorders. The project will randomize participants with depression, anxiety, and/or traumatic stress disorders to one of two doses of cognitive training or a no-treatment control condition. The investigators will examine executive functioning change with cognitive task performance and functional neuroimaging assessments.

ELIGIBILITY:
Inclusion Criteria:

* age 21-55
* fluent in English
* diagnosis of mood, anxiety, or traumatic stress disorder
* clinically elevated repetitive negative thinking
* outpatient status
* 6-week stability if taking selective serotonin reuptake inhibitor (SSRI) medications

Exclusion Criteria:

* past year diagnosis of severe alcohol or moderate or greater substance use disorder
* lifetime history of psychotic or bipolar I disorder
* acute suicidality necessitating immediate clinical intervention
* neurodegenerative or neurodevelopmental disorders
* history of moderate or severe traumatic brain injury or other known neurological condition
* sensory deficits that would preclude completing tasks
* conditions unsafe for completing MRI scanning (e.g., metal in body)
* currently receiving psychosocial treatment
* currently receiving psychiatric pharmacotherapy, except SSRIs

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Repeat Assessment: Repeated assessment only
Period: Overall Study
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
Started | 24 | 24 | 24
Completed | 24 | 18 | 22
Not Completed | 0 | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment | Total
Number analyzed (Participants) | 24 | 24 | 24 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (8.05) | 33.12 (8.93) | 31.59 (7.79) | 31.84 (8.15)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 18 | 17 | 21 | 56
  Male | 5 | 6 | 3 | 14
  Other | 1 | 0 | 0 | 1
  Missing | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 1 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 13 | 16 | 14 | 43
  More than one race | 5 | 2 | 5 | 12
  Unknown or Not Reported | 0 | 5 | 2 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 24 | 24 | 72

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Performance
Description: Span Working Memory Score. Scores are calculated based on memory accuracy total points across all trials, with higher scores indicating better performance (0-81 range).
Time Frame: Baseline, Week 4
Population: Sample reflects missing data for high and repeat assessment groups
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
Number analyzed (Participants) | 24 | 17 | 22
score on a scale | 4.92 (8.07) | 8.18 (14.03) | .27 (10.58)

2. Secondary Outcome: Change in Reading Span Blood Oxygen Level Dependent (BOLD) Response
Description: Functional Magnetic Resonance Imaging (fMRI) Reading span working memory capacity task while undergoing functional MRI. Neural activation to task condition is measured using % signal change (0-100) with higher scores indicating greater activation.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: percent BOLD signal change ROI1
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
Number analyzed (Participants) | 21 | 18 | 18
percent BOLD signal change ROI1 | -2.90 (6.16) | -2.16 (6.62) | 2.46 (3.19)

3. Secondary Outcome: Change in Emotional Working Memory Blood Oxygen Level Dependent (BOLD) Response
Description: Functional Magnetic Resonance Imaging (fMRI) emotional working memory capacity task while undergoing functional MRI. Neural activation to task condition is measured using % signal change (0-100) with higher scores indicating greater activation.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: percent BOLD signal change ROI1
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
Number analyzed (Participants) | 22 | 16 | 16
percent BOLD signal change ROI1 | .21 (1.26) | .58 (1.28) | -1.56 (1.09)

4. Secondary Outcome: Change in Neuropsychological Performance
Description: Change from baseline in neuropsychological performance as measured by the following tests: Flanker Inhibitory Control and Attention Test, Picture Sequence Memory Test, List Sorting Working Memory Test, Oral Reading Recognition Test, Dimensional Change Card Sort Test, Pattern Comparison Processing Speed Test, Matrix Reasoning, Digit Span, Trail Making Test, Digit Symbol Matching, composite score (change in NIH corrected fluid cognition t score) with larger scores reflecting larger gains (1-100 range; T score of 50 is mean with standard deviation of 10).
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
Number analyzed (Participants) | 23 | 17 | 19
T score | 4.35 (6.79) | 7.94 (6.91) | 1.37 (7.67)

5. Secondary Outcome: Anxiety Symptoms
Description: Change from baseline in anxiety symptoms as measured by General Anxiety Disorder 7 (GAD-7). The total score ranges from 0-21. With higher scores indicating higher levels of anxiety symptoms.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
Number analyzed (Participants) | 24 | 18 | 22
score on a scale | -1.21 (4.59) | -4.28 (6.59) | -1.14 (5.78)

6. Secondary Outcome: Symptoms of Depression
Description: Change from baseline in symptoms of depression as measured by the PhenX Depression-Quick Inventory of Depressive Symptoms (QUIDS). The total score ranges from 0-27, with higher scores indicating higher depressive symptoms.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
Number analyzed (Participants) | 24 | 18 | 21
score on a scale | -2.46 (4.77) | -1.56 (5.92) | -1.48 (3.31)

7. Secondary Outcome: PTSD Symptoms
Description: Change from baseline in PTSD symptoms as measured by PTSD Checklist for DSM-5 (PCL-5).The total score ranges from 0-80, with higher scores indicating higher severity.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
Number analyzed (Participants) | 24 | 18 | 22
score on a scale | -6.46 (14.82) | -4.39 (15.32) | -7.91 (10.99)

8. Secondary Outcome: Change Repetitive Negative Thinking (RNT)
Description: Change from baseline in RNT as measured by the Ruminative Response Scale (RRS), Penn State Worry Questionnaire (PSWQ), the Repetitive Negative Thinking Questionnaire-10 (RTQ-10) and the Perseverative Thinking Questionnaire (PTQ) composite z score (z score of 0 reflects mean, larger scores reflecting worse symptoms).
  The total score for the RRS ranges from 22 to 88, with higher scores indicating higher degrees of ruminative symptoms.
  The total score for the PSWQ ranges from 16 to 80, with higher scores indicating higher worry.
  The total score for the RTQ-10 ranges from 10 to 50, with higher scores indicating higher repetitive thinking.
  The total score for the PTQ ranges from 0 to 60, with higher scores indicating higher repetitive negative thinking. Scores of each characteristic of RNT can also be obtained.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: Z score
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
Number analyzed (Participants) | 24 | 18 | 22
Z score | -.09 (.67) | -.12 (.72) | .01 (.80)

9. Secondary Outcome: Self-reported Attention Attention
Description: Change from baseline in attention focusing and attention shifting as measured by the Attention Control Questionnaire. The total score ranges from 20 to 80, with higher scores indicating higher levels of attention control.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
Number analyzed (Participants) | 24 | 18 | 22
score on a scale | -.04 (5.05) | 1.89 (5.30) | 1.05 (3.80)

10. Secondary Outcome: Emotion Regulation
Description: Change from baseline in emotion regulation tendencies as measured by the Emotion Regulation Questionnaire (ERQ). Scores are obtained by averaging the scores of two subscales: cognitive reappraisal and expressive suppression. Higher scores indicating higher use of emotion regulation (10 to 70 range).
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
Number analyzed (Participants) | 24 | 18 | 22
score on a scale | -1.04 (6.96) | -1.06 (8.35) | .59 (7.42)

11. Secondary Outcome: Disability
Description: Change from baseline in disability across six domains, understanding and communicating, getting around, self-care, getting along with people, life activities, and participation in society as measured by the World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0).
  A simple score for the WHODAS 2.0 ranges from 36-180 with higher scores indicating the degree of functional limitations. An item-response-theory based score can also be obtained by summing the recoded item scores within each of the six domains, summing the domains, and converting the summary score into a metric ranging from 0 to 100, with higher scores indicating higher disability.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
Number analyzed (Participants) | 24 | 18 | 22
score on a scale | -1.66 (2.21) | -1.42 (2.14) | -.32 (1.56)

12. Secondary Outcome: Suicide Cognitions
Description: Change from baseline in suicide-related beliefs as measures by the Suicide Cognitions Scale-Revised (SCS-R). The total score ranges from 0 to 64, with higher scores indicating higher severity of suicidal cognitions.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
Number analyzed (Participants) | 24 | 18 | 22
score on a scale | -2.79 (7.67) | -5.44 (10.85) | -5.18 (6.65)

13. Secondary Outcome: Alcohol Use
Description: Change from baseline in drinking patterns as measured by the Alcohol Use Disorders Identification Test (AUDIT). The total score ranges from 0 to 40, with higher scores indicating higher risk. Such that 1-7 indicates low risk, 8-12 risky, and 13+ high risk.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
Number analyzed (Participants) | 24 | 18 | 22
score on a scale | .17 (1.76) | -.17 (1.47) | .14 (2.17)

14. Secondary Outcome: Drug Abuse
Description: Change from baseline in drug abuse as measured by the Drug Abuse Screening Test (DAST-10). The total score ranges from 0-10, with higher scores indicating higher degree of drug abuse related problems.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
Number analyzed (Participants) | 24 | 18 | 22
score on a scale | .00 (.78) | .11 (.76) | -.09 (.81)

15. Secondary Outcome: Insomnia
Description: Changes from baseline in insomnia problems as measured by the Insomnia Severity Index (ISI). The total score ranges 0-21, with higher scores indicating severity of insomnia.
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
Number analyzed (Participants) | 24 | 18 | 22
score on a scale | -.21 (4.38) | -3.06 (5.67) | -2.09 (4.64)

16. Secondary Outcome: Change in Mood and Emotions: Negative Affect
Description: Changes from baseline in mood and emotions as measured by the Positive and Negative Affect Schedule (PANAS).There are two scores calculated, one for positive affect and one for negative affect. The total score for positive affect ranges from 10 to 50. The total score for negative affect ranges from 11 to 55 (higher is greater emotion on the dimension).
Time Frame: Baseline, Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
Number analyzed (Participants) | 24 | 18 | 22
score on a scale | -3.38 (7.14) | -5.06 (9.77) | -.38 (5.07)

17. Secondary Outcome: Change in Mood and Emotion: Positive Affect
Description: as for outcome 16
Time Frame: Baseline, 4 weeks
Population: Reflects missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Repeat Assessment: Repeat assessment group
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
Number analyzed (Participants) | 24 | 18 | 22
score on a scale | 1.25 (13.25) | 2.55 (12.12) | .32 (10.33)

ADVERSE EVENTS:
Time Frame: Baseline through post-treatment assessment (approximately 6 weeks)
Arm/Group | Cognitive Training Low Dose | Cognitive Training High Dose | Repeat Assessment
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT04912089/Prot_SAP_001.pdf
  • Informed Consent Form (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/89/NCT04912089/ICF_000.pdf